CLINICAL TRIAL: NCT02833441
Title: The Peer Support Intervention - Supporting HIV Positive Adolescents in Zimbabwe to Improve HIV Care Continuum Outcomes
Acronym: PESU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zimbabwe (Other)
Responsible Party: Principal Investigator, Azure Tariro Makadzange, Lecturer, University of Zimbabwe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Peer Support Intervention; No. AID-OAA-A-14-00046 (Other: JSI Research & Training Institute, Inc. (JSI))
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer Support Intervention (Experimental): Adolescents/young adults in the Peer Support Intervention arm will be referred to a Peer Support Intervention support group within their own or nearby community. This support group will meet monthly and will be facilitated by a professional HIV counsellor together with a Peer Support Intervention counselor. The Peer Support Intervention counsellors will provide regular counselling to their allocated participants through home visits and SMS messages. Each participant will be visited once a week in their home. Whatsapp messages will be delivered daily to each participant by the Community Adolescent Treatment Supporters. The agreed messages will briefly enquire about the participant's well-being without specifically making reference to HIV or ARVs. In addition, participants' caregivers will be invited to a 3-session intervention to build knowledge, skills and confidence to better support their adolescents.
  Interventions: Behavioral: Peer Support
- Standard of Care Practice (No Intervention): Participants in the standard of care group will receive adherence evaluations and counseling at the clinic as per the current standard of care. Current procedures involve a group counseling session given on Monday morning during which topics are discussed that are relevant to adolescents. In general children aged between 13-19 years attend these sessions. After the group counseling, adolescents also receive an individual counseling session before being evaluated by the clinic doctor. Youth are also encouraged to complete a self reported adherence questionnaire and may periodically undergo pill counts by the clinic counselors.
  The adolescents may belong to peer support groups in their communities, however these activities are not part of the clinic program. No interventions are typically targeted at their caregivers.

INTERVENTIONS:
Behavioral: Peer Support
  Arms: Peer Support Intervention

SUMMARY:
Youth with evidence of virologic failure defined as an HIV VL>400 copies/mL on two consecutive occasions at least 1 month apart will be eligible for enrollment. Youth will be randomized to a community based peer counseling support group or clinic based standard of care, with viral load, and drug monitoring evaluations at 3 month intervals to determine the efficacy of the intervention in improving adherence and virologic suppression.

DETAILED DESCRIPTION:
Title The Peer Support Intervention - supporting HIV positive adolescents in Zimbabwe to improve HIV care continuum outcomes

Short Title The Peer Support Intervention

Study Design Prospective randomized study

Study Duration 2 years

Study Population 250 Youth (ages 10-24 years) with virologic failure

Study Outcomes Primary Outcomes

1. Virologic suppression rate in the The Peer Support Intervention group compared with the standard of care group following 48 weeks in the Peer Support Intervention.

Secondary Outcomes

1. Frequency of acquired drug resistance mutations among youth failing ART.
2. Baseline prevalence of psychological distress among adolescents and young adults failing first line therapy
3. Prevalence of psychological distress (measured using PHQ-A and SSQ) after 48 weeks of enrolment in the Peer Support Intervention compared with the standard of care
4. Association between self-reported adherence, pill counts and objective surrogate markers of adherence obtained from plasma (viral load), DBS and hair (tenofovir concentrations).
5. Effectiveness of point mutation assays for the detection of drug resistance as compared with standard sequencing techniques.

Description of Intervention Youth with evidence of virologic failure defined as an HIV VL>400 copies/mL on two consecutive occasions at least 1 month apart will be eligible for enrollment. Youth will be randomized to a community based peer counseling support group or clinic based standard of care, with viral load, and drug monitoring evaluations at 3 month intervals to determine the efficacy of the intervention in improving adherence and virologic suppression.

Study Sites Parirenyatwa Hospital Family Care Centre

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV positive
* Age > 10 years and ≤ 24 years
* Two consecutive HIV VL>400 copies/mL, at least one month apart
* Residence within 50 km of Harare
* Able to provide written informed consent (age 18 or older) or assent (age <18 years)

Exclusion Criteria:

* Inability to provide informed consent or assent
* Past or current involvement in the Zvandiri Intervention Program

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Actual)
Dates: Start 2016-07; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Virologic suppression rate in the Peer Support Intervention i group compared with the standard of care group following 48 weeks in the Peer Support Intervention. | 2 years
  Virologic suppression

SECONDARY OUTCOMES:
Frequency of acquired drug resistance mutations among youth failing ART. | 2 years
  drug resistance mutations
Baseline prevalence of psychological distress among adolescents and young adults failing first line therapy | 2 years
  psychological distress
Prevalence of psychological distress (measured using PHQ-A and SSQ) after 48 weeks of enrolment in the Peer Support Intervention compared with the standard of care | 2 years
  psychological distress
Association between self-reported adherence, pill counts and objective surrogate markers of adherence obtained from plasma (viral load), DBS and hair (tenofovir concentrations). | 2 years
  (viral load), DBS and hair (tenofovir concentrations).
Effectiveness of point mutation assays for the detection of drug resistance as compared with standard sequencing techniques. | 2 years
  detection of drug resistance

CONTACTS AND LOCATIONS:
Overall Officials: Chiratidzo E Ndhlovu, MBChB, Principal Investigator — University of Zimbabwe College of Health Sciences
Locations (1):
- Parirenyatwa Hospital, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No
Data is readily available and can be obtained following review by MRCZ as required in the consent forms.

REFERENCES:
- [Derived] Mtisi TJ, Kouamou V, Morse GD, Dzinamarira T, Ndhlovu CE. Comparing pill counts and patient self-reports versus DBS tenofovir concentrations as ART adherence measurements with virologic outcomes and HIV drug resistance in a cohort of adolescents and young adults failing ART in Harare, Zimbabwe. J Infect Public Health. 2024 Sep;17(9):102500. doi: 10.1016/j.jiph.2024.102500. Epub 2024 Jul 17. PMID 39173560
- [Derived] Ndhlovu CE, Kouamou V, Nyamayaro P, Dougherty L, Willis N, Ojikutu BO, Makadzange AT. The transient effect of a peer support intervention to improve adherence among adolescents and young adults failing antiretroviral therapy in Harare, Zimbabwe: a randomized control trial. AIDS Res Ther. 2021 Jun 16;18(1):32. doi: 10.1186/s12981-021-00356-w. PMID 34134738